CLINICAL TRIAL: NCT06169033
Title: Radiomics of Intra-abdominal and Subcutaneous Adipose Tissue Predict the Efficacy of Bariatric Surgery (RISABS)
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yuntao Nie, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: CJBariatric002
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Type 2 Diabetes Mellitus; Bariatric Surgery
Keywords: Obesity; Type 2 Diabetes Mellitus; Radiomics; Abdominal adipose; Subcutaneous adipose; Prediction model
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Using radiomics of intra-abdominal and subcutaneous adipose tissue and clinical features to predict the weight loss efficacy and remission of type 2 diabetes mellitus after bariatric surgery.

DETAILED DESCRIPTION:
In this study, the investigator intend to collect abdominal CT from patients who are proposed to undergo bariatric surgery, to extract the radiomics of intra-abdominal fat and subcutaneous fat, and to establish a prediction model for predicting the efficacy of weight loss and remission of type 2 diabetes mellitus at 1 year, 3 years, and 5 years postoperatively, in conjunction with the clinical data.

ELIGIBILITY:
Inclusion Criteria:

* BMI>27.5kg/m2; Type 2 diabetes mellitus; Patients who will undergo bariatric surgery

Exclusion Criteria:

* Patients without abdominal CT scan; Patients did not undergo sleeve gastrectomy or Roux-en-Y gastric bypass.

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Obese patients with type 2 diabetes who will undergo bariatric surgery (sleeve gastrectomy or Roux-en-Y gastric bypass) and receive abdominal CT scan will be included in the study.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) of the weight loss prediction model after 1 year | 1 year
  This metric shows the discriminatory ability of the radiomic model to predict the probability of inadequate weight loss after 1 year.
Area under curve (AUC) of the T2DM remission prediction model after 1 year | 1 year
  This metric shows the discriminatory ability of the radiomic model to predict the probability of remission of T2DM after 1 year.

SECONDARY OUTCOMES:
Area under curve (AUC) of the weight loss prediction model after 3 years | 3 years
  This metric shows the discriminatory ability of the radiomic model to predict the probability of inadequate weight loss after 3 years.
Area under curve (AUC) of the T2DM remission prediction model after 3 years | 3 years
  This metric shows the discriminatory ability of the radiomic model to predict the probability of remission of T2DM after 3 years.
Area under curve (AUC) of the weight loss prediction model after 5 years | 5 years
  This metric shows the discriminatory ability of the radiomic model to predict the probability of inadequate weight loss after 5 years.
Area under curve (AUC) of the T2DM remission prediction model after 5 years | 5 years
  This metric shows the discriminatory ability of the radiomic model to predict the probability of remission of T2DM after 5 years.
Area under curve (AUC) of the weight regain model | 5 years
  This metric shows the discriminatory ability of the radiomic model to predict the probability of weight regain.
Area under curve (AUC) of the T2DM relapse model | 5 years
  This metric shows the discriminatory ability of the radiomic model to predict the probability of T2DM relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Nie, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Yuntao Nie, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Subject information involves medical and personal privacy and access is subject to the consent of the principal investigator.